CLINICAL TRIAL: NCT00963352
Title: Prognosis of Colon Cancer. Clinical and Pathological-anatomical Factors Concerned With Radical Surgery
Brief Title: Colon Cancer Prognosis After Radical Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haraldsplass Deaconess Hospital (Other)
Responsible Party: Karl Sondenaa, professor, University of Bergen, Haraldsplass Deaconal Hospital, Department of Surgery, Bergen, Norway
Other Study IDs: Knut2009
Record Dates: First submitted 2009-08-19; First posted 2009-08-21 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Colon Cancer
Keywords: Colon cancer; Open surgery resection; Laparoscopic surgery resection; Morbidity; Mortality; Metastases; Oncology; Freedom of malignant disease recurrence; Safety of intervention open and laparoscopic; Examination of adverse markers; Development of metastases in lungs and other organs
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies. 1) fresh frozen 2) sampled in RNA later 3) archival formalin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients operated for colon cancer

SUMMARY:
1. Radical surgery. It is supposed to improve prognosis of colon cancer. A surrogate measure of achievement of radical surgery is the number of lymph nodes removed with the specimen.
2. Markers. There may be variables that may make patient assessment more sound. The project is including investigation of such markers (genes, old age, comorbidity, and others).
3. Laparoscopic resections. This is being used more and more in cancer surgery but the feasibility of this approach remains to be proven compared with conventional open surgery. The project compares these according to 1) and 2).
4. Morbidity and mortality must be surveilled to keep at a minimum. Many patients have comorbidity and are old to make this factor extra important, including perioperative care.
5. Proper treatment of colon metastases may prolong life. Treatment of lung-metastases will be studied in particular.

DETAILED DESCRIPTION:
1. Radical surgery. A detailed description of procedures for each location of tumor in the large intestine is used. By following a given procedure for each location in the large intestine, the number of lymph nodes can be analyzed for each location to find out if this differs and if prognosis is affected by lymph node numbers according to tumor site.
2. Markers. Different variables are examined for use in clinical judgment to make treatment better as well as genetic experimental analyses for comparison with clinical outcome to better understanding of clinical behavior.
3. Laparoscopic resections. The technical challenge of laparoscopic approach has been compared with conventional surgery without any difference being observed in trials. However, it should be compared with radical open surgery to compare best achievements by using number of lymph nodes as well as outcome measures in the short and long term (mortality).
4. Comorbidity, old age itself, type of surgery and perioperative care according to the so called fast track surgery may all play a part in reducing perioperative morbidity and mortality. A maximum 3% mortality should be aimed for.
5. Colon cancer usually metastasize to the liver and lungs. Surgical treatment of liver metastases has been extensively studied and the prognosis has improved. Lung metastases has not been given similar attention but the prognosis of those operated may be good and equal that after liver surgery. The need for pulmonary resection and factors associated with metastases and lung metastases in particular will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Malignant tumor (adenocarcinoma) of the large intestine (colon)
* Willingness to participate

Exclusion Criteria:

* No radical resection (R0) possible
* Unwilling to participate or medically unfit to undergo follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community patient population from hospital catchment area.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival (DFS) | 2007/10 - 2010/13

SECONDARY OUTCOMES:
5-year overall survival (OS) | 2007/10 - 2012/15

CONTACTS AND LOCATIONS:
Overall Officials: Karl Sondenaa, MD, PhD, Study Chair — Haraldsplass Deaconal Hospital, University of Bergen, Norway
Locations (2):
- Norway (2):
  - Haraldsplass Deaconal Hospital, Department of Surgery, Bergen
  - Haukeland University Hospital, Bergen